CLINICAL TRIAL: NCT03009253
Title: Translational Research on Locally Advanced Pancreatic Adenocarcinoma
Acronym: TRLAPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Chengfeng Wang, Director of department of pancreatic and gastric surgery, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GHGI061
Record Dates: First submitted 2016-12-22; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Pancreatic Cancer
Keywords: Neoadjuvant therapy; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concurrent chemoradiotherapy(CCRT) Group (Experimental): Concurrent chemoradiotherapy (Total dose: 30-40 Gy; Single dose: 3-4 Gy; Frequency: 10; S-1 orally (80 mg/m2/d),2 weeks) Followed by chemotherapy: Gemcitabine(GEM), 1000 mg/m2 ,Day 1,8 ); taking S-1 orally (80 mg/m2/d, bid on Day 1-14, Q21d, 3 cycles)
  Interventions: Other: order of treatment
- Chemotherapy Group (Experimental): Chemotherapy (Gemcitabine(GEM), 1000 mg/m2 ,Day 1,8 ); taking S-1 orally (80 mg/m2/d, bid on Day 1-14, Q21d, 3 cycles)
  Followed by Concurrent chemoradiotherapy:
  (Total dose: 30-40 Gy; Single dose: 3-4 Gy; Frequency: 10; S-1 orally (80 mg/m2/d),2 weeks)
  Interventions: Other: order of treatment

INTERVENTIONS:
Other: order of treatment — the 2 arms have different orders of treatment,participants in arm A accept concurrent chemoradiotherapy at first and then accept evalution for surgery.In arm B,participants accept concurrent chemoradiotherapy at first and then accept evalution for surgery.

SUMMARY:
The purpose of this study is to find the best neoadjuvant therapy for pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
The trial is prepared to be registered on the clinicaltrail.gov. Quality assurance plan: Every participant is enrolled or excluded by two practiced investigators. And two investigators participated in all steps of the trail, including the record of the data, and the investigators will compare the data. If the data is consistent,the investigators would record the data; if not, the data would be checked and decided by the two investigators. All the steps and data are site monitored and audited by the workers of research and financial department of National Cancer Center/ Cancer Hospital, Chinese Academy of Medical Sciences.

Data check: The investigators compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources, including medical records and electronic case report forms.

Data dictionary that contains detailed descriptions of each variable used by the registry,including the source of the variable, coding information, and normal ranges if relevant.Standard Operating Procedures to address registry operations and analysis activities,such as participants recruitment, data collection, data management, data analysis,reporting for adverse events, and change management. All registry operations would be done according to specific steps, and by two practiced investigators.

Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect. According to the formula to differ advantages and disadvantages, the investigators need at least 80 participants to take part in the trail.

The investigators can recruit about 20 participants every year according to previous experiences, so the investigators should recruit at least for two years.

Plan for missing data: the investigators would collect as much data as possible, and the investigators exclude the participants who cannot cooperate on recruitment. And the investigators manage situations according to statistical principles where variables are reported as missing, unavailable, "non-reported," uninterpretable, or considered missing because of data inconsistency or out-of-range results.

Statistical analysis plan: Kaplan-Meier method would be used to analyze the difference of survival time between the two groups, and the local control rate of the two groups would be compared by chi square test. Statistical analyses would be performed by using IBM SPSS Statistics(version 20; IBM, Chicago, USA). The level of significance is defined as P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* have cytologic or pathological proof of pancreatic adenocarcinoma without surgery contraindication score of ECOG is between 0 and 1 evaluation of CT is unresectable

Exclusion Criteria:

* metastatic pancreatc adenocarcinoma malignant tumors history allergic to 5-FU have difficulty in swallowing joined other clinical trails cardiac and renal disease active infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
translational resection rate | half a year

SECONDARY OUTCOMES:
progression-free survival | 2 years
  PFS
Local control rate | 2 years
  LCR

CONTACTS AND LOCATIONS:
Overall Officials: Chengfeng Wang, B.A., Principal Investigator — Investigator CancerIHCAMS
Locations (1):
- Cancer Institute and Hospital ,China Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided